CLINICAL TRIAL: NCT02332642
Title: Immuno-monitoring of Patients With Metastatic Melanoma (AJCC Stadium IV) Under Chemotherapy
Acronym: ImmunoPAX
Status: Completed | Type: Observational
Sponsor: Universitätsmedizin Mannheim (Other)
Responsible Party: Principal Investigator, Dr. Christoffer Gebhardt, Principal Investigator, Universitätsmedizin Mannheim
Other Study IDs: 2014-624N-MA
Record Dates: First submitted 2015-01-05; First posted 2015-01-07 (Estimated); Last update posted 2017-03-07 (Actual); Status verified 2017-03

CONDITIONS: Immuno-monitoring

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Immuno-monitoring

SUMMARY:
This pilot clinical trial aims at evaluating immuno-modulating effects of palliative treatment with specifically dosed standard chemotherapeutics in patients with metastatic melanoma (AJCC stage IV) by assessing myeloid-derived suppressor cells' (MDSCs) count and activity.

ELIGIBILITY:
Inclusion Criteria:

* histologically defined metastatic melanoma patients (AJCC stage IV)
* aged 18 to 80 years
* at least one prior systemic anti-melanoma therapy; if BRAFV600 positive, at least one prior BRAFi therapy

Exclusion Criteria:

* therapy-naive patients
* any contra-indications for (specific) systemic chemotherapy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Metastatic melanoma patients (AJCC stage IV)
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2014-11; Primary Completion 2016-12 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Immuno-monitoring | Immediate

CONTACTS AND LOCATIONS:
Overall Officials: Christoffer Gebhardt, M.D., Principal Investigator — Universitätsmedizin Mannheim; Jochen Utikal, M.D., Principal Investigator — Universitätsmedizin Mannheim
Locations (1):
- Universitätsmedizin Mannheim, Klinik für Dermatologie, Venerologie und Allergologie, Mannheim, Germany

REFERENCES:
- See also: Homepage — http://www.dkfz.de/en/dermato_onko/index.php